CLINICAL TRIAL: NCT01722786
Title: Prospective, Observational, Non-interventional Open-label Multicenter Registry Regarding the Management of Severe Bleeding and/or Urgent Interventions During Treatment With Direct Oral Anticoagulants or Vitamin K Antagonists
Brief Title: Reversal Agent Use in Patients Treated With Direct Oral Anticoagulants or Vitamin K Antagonists
Acronym: RADOA
Status: Completed | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); University Hospital Greifswald (Other); University Hospital Dresden (Other); University Hospital, Aachen (Other); Goethe University (Other); University Hospital Schleswig-Holstein (Other); Vivantes Netzwerk für Gesundheit GmbH (Other); Ruhr University of Bochum (Other); Technische Universität Dresden (Other); Städtisches Klinikum Dresden-Friedrichstadt (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. E. Lindhoff-Last, M.D., Cardioangiologisches Centrum Bethanien
Other Study IDs: RADOA-Registry
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Severe Bleeding; Urgent Surgery
Keywords: severe bleeding; dabigatran; rivaroxaban; apixaban; edoxaban; PCC; aPCC; rVIIa; hemodialysis; antidots; idarucizumab
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — If possible, left-over from plasma samples ("retention sample") should be used to perform further analyses as drug concentrations. Retention samples of very low volume would suffice for HPLC (information on collection method needed) to assess plasma concentrations of anticoagulants in these patients.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- DOA: Expected number of patients estimated by study duration
  N= 90 patients treated with direct oral anticoagulants (DOA) with acute bleeding
  N= 40 patients treated with direct oral anticoagulants (DOA) with urgent surgical intervention
- VKA: Expected number of patients estimated by study duration
  N= 90 treated with vitamin K antagonists (VKA) with acute bleeding
  N= 40 patients treated with vitamin K antagonists (VKA) with urgent surgical intervention

SUMMARY:
Patients treated with Vitamin K antagonists (VKA) or direct oral anticoagulants as Rivaroxaban, Apixaban, Edoxaban or Dabigatran, who experience severe bleeding and/or need urgent interventions/operations that cannot wait are included in this registry, or during emergency operations.

DETAILED DESCRIPTION:
The Registry will offer the opportunity to evaluate the effects of reversal agents as PCC, aPCC, rVIIa, specific antidots in e.g. severe bleeding patients treated with oral anticoagulants.

By collecting case reports from several university hospitals and clinics, different treatment strategies in clinical practice will be observed and evaluated, and may serve as a comprehensive information resource for the safe management with DOA, but also with the long-term anticoagulation based on coumarin derivatives in the near future.

The current objective of this registry is to:

1. Document the clinical course and outcome of various clinical bleeding events associated with DOA or VKA in patients with severe life-threatening bleeding making intervention necessary
2. Document the clinical course and outcome of urgent surgical interventions within 24 hours after admission in patients under DOA or VKA treatment.
3. Characterisation of therapeutic strategies in stopping acute life-threatening bleeding including following agents and methods:

   1. blood transfusion,
   2. platelet concentrates
   3. reversal agents [e.g. vitamin K, prothrombin complex concentrate (PCC), activated PCC (aPCC), activated factor VII (aVII), fibrinogen concentrate, fresh frozen plasma (FFP)]
   4. specific antidots, e.g. idarucizumab
   5. haemodialysis
   6. desmopressin
   7. tranexamic acid
   8. no specific treatment in respect to the above mentioned treatments (e.g. stop of medication and waiting until anticoagulant effect of DOA is decreased).

ELIGIBILITY:
Patient Eligibility

1. a) Bleeding patients:

   Anticoagulated patients with DOA or VKA with clinically overt major bleeding according to a specified ISTH definition for non-surgical patients:
   * Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome
   * Bleeding causing a fall in hemoglobin level of 2 g L-1 (1.24 mmol L-1 ) or more leading to transfusion of two or more units of whole blood or red cells.

   OR b) Acute surgical need Patients treated with DOA or VKA and who need urgent operation which cannot wait (< 24 h after last intake of drug)

   AND
2. with or without reversal agent use (e.g. PCC, aPCC, rVIIa) (and/or haemodialysis for dabigatran)

   AND
3. provides informed consent after the acute event

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Expected number of patients estimated by study duration
  N= 90 patients treated with direct oral anticoagulants (DOA) with acute bleeding N= 90 treated with vitamin K antagonists (VKA) with acute bleeding
  N= 40 patients treated with direct oral anticoagulants (DOA) with urgent surgical intervention N= 40 patients treated with vitamin K antagonists (VKA) with urgent surgical intervention
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2014-04; Primary Completion 2018-06-30 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | open
  Primary observation points (for all patients):
  In hospital mortality up to 30 days after admission
  Secondary observation points (group of patients with life threatening bleeding under oral anticoagulation)
  1. Stop of bleeding defined according to the treating physicians
  2. Fatality rate caused by unstoppable bleeding
  3. Use versus no use of reversal agents - difference in outcome?
  4. Definition of supportive measures being effective in stopping bleeding
  5. Effectiveness of specific antidots
  6. Effectiveness of dialysis vs. no dialysis in case of dabigatran accumulation associated with bleeding
  7. Causality assessment: Relation of SAE to anticoagulant medication

SECONDARY OUTCOMES:
Secondary Outcome | open
  Secondary observation points (group of patients with acute surgery under oral anticoagulation)
  1. Blood loss, number of transfusions necessary
  2. Satisfaction of surgeon during and after surgery concerning bleeding
  3. Use versus no use of reversal agents - difference in blood loss and number of transfusions?
  4. Use versus no use of reversal agents - difference in satisfaction of surgeon using a standardized questionnaire
  5. Causality assessment: Relation of SAE to anticoagulant medication
  6. Delay in performance of surgery due to anticoagulation

CONTACTS AND LOCATIONS:
Locations (1):
- Cardioangiology Center Bethanien (CCB), Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindhoff-Last E, Herrmann E, Lindau S, Konstantinides S, Grottke O, Nowak-Goettl U, Lucks J, Zydek B, Heymann CV, Birschmann I, Sumnig A, Beyer-Westendorf J, Schellong S, Meybohm P, Greinacher A. Severe Hemorrhage Associated With Oral Anticoagulants. Dtsch Arztebl Int. 2020 May 1;117(18):312-319. doi: 10.3238/arztebl.2020.0312. PMID 32605708
- [Derived] Pfeilschifter W, Lindhoff-Last E, Alhashim A, Zydek B, Lindau S, Konstantinides S, Grottke O, Nowak-Gottl U, von Heymann C, Birschmann I, Beyer-Westendorf J, Meybohm P, Greinacher A, Herrmann E; RADOA-Registry Investigators (Reversal Agent use in patients treated with Direct Oral Anticoagulants or vitamin K antagonists Registry). Intracranial bleeding under vitamin K antagonists or direct oral anticoagulants: results of the RADOA registry. Neurol Res Pract. 2022 May 2;4(1):16. doi: 10.1186/s42466-022-00183-y. PMID 35491419